



# SIMPLIFIED PROTOCOL RESEARCH NOT INVOLVING THE HUMAN BEING

| TITLE | Real life data from hypertensive patients treated with renal denervation in current practice in France- French RENal Denervation registry |
|---|---|
| SHORT TITLE | FRIEND |
| ORGANISATION RESPONSIBLE FOR THE PROCESSING OF DATA SCIENTIFIC RESEARCH AND IMPLEMENTATION COORDINATORS | CHU GRENOBLE ALPES Courriel: DRCI@chu-grenoble.fr Téléphone: 04 76 76 59.57 Adresse: CS 10217, 38043 Grenoble Cedex 09 Pays: FRANCE Dr Romain Boulestreau Cardiologist Cardiology Department University Hospital Center, Bordeaux email: Romain.boulestreau@chu-bordeaux.fr Phone: 05-56-79-56-79 Address: Hôpital Haut Leveque av Magellan, 33600 Pessac Pr Olivier Ormezzano Cardiologist Hypertension and atherothrombosis University Hospital, Michallon, Grenoble, France |
| LIST OF ASSOCIATED CENTERS | email: oormezzano@chu-grenoble.fr Phone: 04-76-76-88-88 Address: CS 10217 - 38043 Grenoble cedex 09 7 test centers initially (will be extended to 20 centres in a second phase) - Centre n°1: CHU Grenoble Alpes: Pr ORMEZZANO, oormezzano@chu-grenoble.fr, Cardiology department, University Hospital, Michallon CS 10217 - 38043 Grenoble cedex 09 - Centre /Partenaire n°2: Dr DOUBLET, julien.doublet@chu-bordeaux.fr, Cardiology department, Hôpital Haut-Levèque CHU Bordeaux 1 rue Jean Burguet, 33000 Bordeaux-Principal investigator - Centre /Partenaire n°3: Pr AZIZI michel.azizi@aphp.fr Cardiology department, Hôpital Européen Georges-Pompidou HEGP |



20 rue Leblanc. 75015 Paris- Principal investigator Centre /Partenaire n°4: Pr COURAND pierre-yves.courand@chu-lyon.fr Cardiology department 103 GdR Croix Rousse, 69004 Lyon Principal investigator Centre /Partenaire n°5 : Pr DUNY BOUHANIC Hypertension and Therapeutics Department duly-bouhanick.b@chu-toulouse.fr Hôpital Rangueil, 1, avenue du Professeur Jean Poulhès - TSA 50032 - 31059 Toulouse cedex 9 Principal investigator Centre /Partenaire n°6: Dr DELARCHE nicolas.delarche@ch-pau.fr Cardiology department Hospital center, 4 Boulevard Hauterive- 64000 PAU Principal investigator Centre /Partenaire n°7: Dr SILHOL Francois.SILHOL@ap-hm.fr Cardiology department Hôpital de la Timone, 264 rue Saint-Pierre 13385 Marseille Principal investigator Renal denervation (RDN) is a recent procedure that can be used to control BP (blood pressure) in hypertensive patients. Numerous publications from randomised trials have demonstrated the efficacy of RDN in this indication (1-14). The latest guidelines now include RDN as an effective technique for use in hypertension. Since the beginning of 2023, RDN using Medtronic's Spiral radiofrequency system has benefited from transitional authorisation for reimbursement by the French health insurance system. An application for reimbursement is underway for the ultrasound system. We aim to compile an exhaustive prospective register of all procedures BACKGROUND carried out in France over the next few years, regardless of the type of catheter used or the context in which the procedure was carried out (transitional reimbursement, industrial register, randomised trial). Our aim is to assess the efficacy and safety of the procedure within the French healthcare system, the characteristics of patients benefiting from the procedure, the centres performing renal denervation, and the care pathways used, and to be able to present all this data, independently of the industry, to the healthcare authorities when it comes time to reassess the value of this procedure and its indications.



| version 12.0 of the protocol model RNIPH | TRIEND registry |
|---|---|
| | □ Diagnostics |
| | ☐ Prevention and treatment |
| | ☐ Patient management |
| | ☐ Patient safety |
| | ☐ Organization of healthcare facilities |
| PRIMARY OBJECTIVE | ☐ Public health policies |
| | ☐ Understanding diseases |
| | ☐ |
| | Measurement (HBPM) in hypertensive patients between before and 1 year after |
| | treatment with RDN. |
| _ | |
| PRIMARY ENDPOINT | Change in SBP measured by HBPM before and after RDN (1 year). |
| | SECONDARY OBJECTIVES: |
| | - To evaluate changes in office systolic blood pressure, the combination of SBP measured in HBPM and day ABPM and 24-hour SBP before and 3 months, 6 |
| | months, 1 year, after DNR. |
| | - Evaluate the evolution at 3 months, 6 months, 1 year, of the drug burden in |
| | antihypertensive treatment (DDD), the percentage of patients having reached the blood pressure target and the win ratio. |
| | - Evaluate the development of renal artery stenosis before and 6 months, 1 year, |
| | after DNR Evaluate the evolution of creatinine levels before and 6 months, 1 year, after |
| SECONDARY OBJECTIVES | DNR. |
| | - Evaluate the occurrence of other complications related to hypertension or to the procedure itself. |
| | - Comparison of responders and non-responders to the procedure (24h ABPM |
| | systolic blood pressure decrease of 5 mmHg or more and/or the diminution of the medical burden by at least one therapeutic class without SBP increase compared |
| | to baseline). |
| | - Evaluate the performance of known predictors of response to renal denervation |
| | <ul><li>in our population.</li><li>- Describe the type of center performing the procedure, the context in which DNR</li></ul> |
| | is performed, patient characteristics and care pathways. |
| METHODOLOGY | Research that does not involve the human person, as it involves the prospective, retrospective, descriptive and comparative use of multicentric data from routine |
| | care. |
| TYPE OF DATA COLLECTED | The data collected are detailed below: |
| | Administrative data: |
| | - centre number followed by a hyphen (-) then the patient's number |
| | - collection of the patient's non-objection to participate in the FRiEND register - date of inclusion, date of procedure |
| | aute of inclusion, dute of procedure |



- type of centre carrying out the procedure (hospital, university hospital, clinic, ESPIC, other)
- setting in which the procedure was carried out (day hospitalisation, week hospitalisation, conventional hospitalisation)

#### • Personal data:

- Patient's initials, date of birth (in MM/YYYY format).
- Gender (male, female, not gendered, refuses to answer), height, weight,

## • Biological data:

- Biological work-up with measurement of the following parameters: Plasma ionogram (Na, K), blood count and platelet count (NFP), proteinuria, fasting glycaemia, total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, creatininaemia, estimated glomerular filtration rate (eDFG) (according to the Modification of Diet in Renal Disease (MDRD) method), uricaemia, microalbuminuria or urinary albumin/creatinine (assessment of target organ damage).

#### • Clinical data:

- Systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR): three measurements will be taken with a validated oscillometric electronic device measured according to international recommendations (2023ESH-ESC)
- risk factors (dyslipidaemia, type 2 diabetes, hypertension, smoking)
- cardiovascular (CV) history of more than 6 months (myocardial infarction, coronary insufficiency, stroke)
- non-CV history (cancer, asthma or respiratory insufficiency, musculoskeletal disability)
- ABPM measurement (SBP and DBP for 24 hours, during the day and at night)
- self-measurement of BP (according to the rule of 3 : average of 3 measurements in the morning and 3 in the evening, 3 consecutive days).
- current treatments (anti-hypertensive, lipid-lowering, anti-diabetic, anti-platelet).
- Therapeutic adherence assessment

## • Imaging data:

- results of CT scan of renal arteries: number of renal arteries, diameter of renal arteries, assessment of possible renal artery stenosis (in %)
- Renal artery echodoppler (if feasible): assessment of possible renal artery stenosis (in %), renal artery blood flow velocity.

CHU

Version n° 1.0 du 03/04/2025

#### Procedure:

- Indication validated by a Centre of Excellence or Blood Pressure Clinic (yes/no)
- Complete secondary hypertension work-up (yes/no)
- In particular: plasma renin/aldosterone assay? Methoxylated catecholamine derivatives? renal artery imaging?
- Precise indication of the procedure
- context of treatment (temporary reimbursement of SIMPLICITY catheters, registry, randomised study)
- specialities of the doctor(s) performing the procedure,
- details of the procedure: under general anaesthetic/analgesia, approach,
- Antithrombotics and anti-platelet aggregants before, during and after the procedure
- number of ablation/sonication points performed
- volume of contrast medium used, X-ray dosimetry
- closure system for the approach port
- complications, if any

### Follow-up data :

- Date and type of follow-up
- Progress of treatment
- clinical BP measurements, MAPA and self-measurements performed
- Changes in biological markers
- Changes in imaging of the renal arteries
- Complications, if any

This might include retrospective data for patients treated with RDN in the past, if investigator believe that the missing data are absent or scarce. As we will collect only data coming from a routine care already widely used in France for these patients, this should correspond to most of the patients already treated with RDN. Patients included retrospectively and prospectively will be compared to ensure that there are no selection biaises in the retrospective cohort.

Use one or more of the following sensitive variables:

☐ Country and department of residence of the person studied (NB: the

collection of the commune of residence (zip code and/or name) is not permitted)

Pays et département de résidence de la personne étudiée (NB : le recueil de la commune de résidence (code postal et/ou nom) n'est pas autorisé)

☑ Year and month of birth



| | ☐ Date of care (DDMMYYYY) |
|---|---|
| | ☐ Date of death (DDMMYYYY) ☐ City of death |
| | □ None |
| | ⊠Medical record |
| | ☐ Survey / Cohort / Register not including SNDS data |
| ORIGIN OF DATA | ☐ Other data |
| ORIGIN OF DATA | <ul> <li>☑ Data from the investigator's department only (coordinating and associated centers)</li> <li>☐ Data from several departments of the CHU Grenoble Alpes or from a</li> </ul> |
| | department other than that of the investigator (if the investigator is at no time |
| | involved in the care of the persons targeted by the research). Prospective and restrospective research: |
| DATA COLLECTION SCHEDULE | <ul> <li>3-year register (start of collection april 2025 - end of inclusions april 2027, follow-up: 1 year)</li> <li>For retrospective patients, data collection will be done from clinical database from january 2010. A 4-week delay must be observed between the sending of information letters and the start of data collection.</li> <li>End of follow-up: april 2028.</li> <li>Annual analysis of data from patients who have undergone RDN and follow-up at 1 month, 6 months, 1 year after the procedure.</li> </ul> |
| DATA COLLECTION | Collection: The data collected will be those from routine follow-up at 1 month, 6 months, 1 year of all patients benefiting from a RDN procedure and included in the registry. After the procedure, the investigator in each participating centre will manage the follow up of the patient. As the study is purely observational, it does not require any specific follow-up visits, but includes the collection of data obtained during routine follow-up visits. The registry does, however, include data collection at fixed times after procedure. The data reported in the Redcap file will be the data available closest to the theoretical day of collection. Patients who have been lost to follow-up should be investigated through the referring doctors to RDN and/or by family members or any other person whose name appears on the patient liaison form. In the absence of any information, a search for the patient's possible death will be carried out by consulting the https://deces.matchid.io/searchqui website, including the INSEE source for deaths (the search will be carried out by birth name). In case of of the patient's death, the medical record is first checked to ensure that the patient has "no objection" to the use of his or her health data for research purposes. Clinical data collection will be based on the source documents. |



| Version 12.0 of the protocol model RNIPH | FRIEND registry | Version n° <b>1.</b> 0 du 03/04/2025 |
|---|---|---|
| | Codage: The data will be pseudonymised by coding: patients will be identified. | |
| | follows: centre number followed by a hyphen (-) then the patient numb | |
| | coded number specific to the research indicating the order of inclusion | |
| | subjects (ex. 01-001). The list of correspondences between the patient cod | |
| | and his identity will be kept in each participating center, in the servic | |
| | server, by the investigator on an Excel file. | |
| DATA STORAGE PERIOD | Personal data relating to persons taking part in resepurpose, may be kept in the information systems of the centre or the healthcare professional involved in the years after the last publication of the results of the publication, until the final report of the research is since The personal data of the professionals involved in the formore than fifteen years after the end of the last reparticipated. It is then archived on paper or electronically for a with the regulations in force. The data must then be | ne controller, the participating research for a maximum of 2 ne research or, if there is no igned. the research may not be kept esearch project in which they period of time in accordance |
| | NUMBER OF SUBJECTS TO BE INCLUDED | |
| | The number of subjects included will correspond undergoing renal denervation for hypertension a Hospital and in the various French centres particip study period (the estimation is currently 100 per year | at the Grenoble University ating in the study during the |
| DESCRIPTION OF<br>STATISTICAL ANALYSIS<br>OF DATA | DATA ANALYSIS The database will be stored in accordance we commitment, on a secure database certified to keep REDCAP system supporting the eCRF. The analyst University Cardiology Clinic of the Grenoble University Cardiology Clinic Oniversity Cardi | health data, and linked to the<br>ses will be carried out at the<br>versity Hospital by Professor<br>he help of the SFHTA, using |
| | Statistical analysis: Absolute values, percentages calculated to describe the population. The differences between the variables before and a using either a paired t-test for normally distributed of paired Chi2 or a Fisher test. For univariate analysis of responder groups (5 mmHg reduction in 24h SBP) use the t-student analysis of variance test or non-pa variables, and chi2 or Fisher tests for categorical variables be performed. | after the RDN will be tested data or a Wilcoxon test, and a of variables between the RDN and non-responders, we will arametric tests for continuous ables. A multivariate analysis |
| | Number of subjects: Estimation of 100 per year (n | |
| PEOPLE INCLUDED IN THE | then more as RDN implementation in France increas | se) |
| RESEARCH | Inclusion criteria: Adult (> 18 years old) hypertens. | ive patients treated with RDN |
| | in France whatever the catheter and the indicate | cation. This might include |
| | retrospective data for patient already treated with RI | ON in the past. |



| | Non-inclusion criteria: RDN not proposed to the patient, patient opposing the |
|---|---|
| | collection and use of his/her data for research purposes. |
| | Information and traceability procedures for non-objection/opposition: |
| | Patients will be fully and fairly informed, in comprehensible terms, of the |
| | objectives of the study and the nature of the information collected, and of their |
| | right to object at any time to the use of the data collected. They will be given an |
| | information letter and the non opposition will be written down in the medical |
| | records of the patient. If the subject objects to their personal health data being |
| | processed for research purposes, this objection will be recorded in their medical |
| | file. This right of objection may be exercised at any time by any means with either |
| | the person responsible for the research or the establishment holding the data, |
| | which undertake to respond to the request within a maximum of 2 months. |
| | Retrospective patients will be informed by post. On receipt of this letter, the |
| | patient will have 4 weeks to object. |
| ETHICS | |
| | NA |
| | The legal basis for this data processing is Article 6 of the General Data Protection |
| | Regulation (GDPR), namely the performance of a mission of public interest |
| WHY THE STUDY IS IN | assigned to the data controller and the legitimate interests pursued by it. In |
| THE PUBLIC INTEREST | addition, under Article 9 of the GDPR the data controller may exceptionally |
| | process special categories of data, including health data notably for scientific |
| | research purposes. |
| | To objectively evaluate RDN performance, patients and center profiles and care |
| | pathway in the various French centres participating to the registry, and to |
| | investigate whether there are any predictive factors (on the basis of the initial |
| EVDECTED DEMERITS | clinical and biological work-up) for the outcome in terms of lowering blood |
| EXPECTED BENEFITS | pressure, in order to better target patients who could benefit from this type of |
| | procedure in the future. |
| | Provide informed, independent data to the health authorities to support |
| | reimbursement decisions and the choice of indications. |

 $Version \ 12.0 \ of \ the \ protocol \ model \ RNIPH \\ FRIEND \ registry \\ Version \ n^{\circ} \ \textbf{1.0} \ du \ 03/04/2025$ 

# Study schedule

| Visits | During | 1 month | 6 | 12 |
|---|---|---|---|---|
| | hospitalization for | after | months | months |
| | RDN | RDN | after | after |
| | | | RDN | RDN |
| Patient information | X | | | |
| RDN indication verification | X | | | |
| Blood sample | X | | | |
| Imaging examinations | X | | | |
| Medical history collection | X | | | |
| Clinical examination | X | X | X | X |
| Ongoing therapy collection | X | X | X | X |
| Adverses events recording | X | X | X | X |
| Blood Pressure and heart rate | X | X | X | X |
| recording | A | Λ | Λ | Λ |
| Blood sample | | | | |
| Ionogram (Na, K), glucose level, | | | | |
| creatininemia (DFG MDRD), | X | X | X | X |
| uricemia | | | | |
| Total Cholestérol, HDL, LDL | | | | |
| triglycerides, NFP | | | | X |
| Microalbuminuria, proteinuria | | | | X |
| Clinical examinations | | | | |
| Home Blood Pressure | | X | X | X |
| Measurement | | | 11 | |
| Ambulatory Blood Pressure | | | | X |
| Measurement | | | | 71 |
| Renal Arteries ultrasound | | | | X |
| Renal arteries angioCT | | | | X |
| | | • | • | |

## Bibliographie:

1. Adherence to Antihypertensive Treatment and the Blood Pressure-Lowering Effects of Renal Denervation in the Renal Denervation for Hypertension (DENERHTN) Trial. Azizi M, Pereira H, Hamdidouche I, Gosse P, Monge M, Bobrie G, Delsart P, Mounier-Véhier C, Courand PY, Lantelme P, Denolle T, Dourmap-Collas C, Girerd X, Michel Halimi J,



Zannad F, Ormezzano O, Vaïsse B, Herpin D, Ribstein J, Chamontin B, Mourad JJ, Ferrari E, Plouin PF, Jullien V, Sapoval M, Chatellier G; DENERHTN Investigators. Circulation. 2016 Sep 20;134(12):847-57.

- 2. Optimum and stepped care standardised antihypertensive treatment with or without renal denervation for resistant hypertension (DENERHTN): a multicentre, open-label, randomised controlled trial. Azizi M, Sapoval M, Gosse P, Monge M, Bobrie G, Delsart P, Midulla M, Mounier-Véhier C, Courand PY, Lantelme P, Denolle T, Dourmap-Collas C, Trillaud H, Pereira H, Plouin PF, Chatellier G; Renal Denervation for Hypertension (DENERHTN) investigators. Lancet. 2015 May 16;385(9981):1957-65
- 3. Abdominal Aortic Calcifications Influences the Systemic and Renal Hemodynamic Response to Renal Denervation in the DENERHTN (Renal Denervation for Hypertension) Trial. Courand PY, Pereira H, Del Giudice C, Gosse P, Monge M, Bobrie G, Delsart P, Mounier-Vehier C, Lantelme P, Denolle T, Dourmap C, Halimi JM, Girerd X, Rossignol P, Zannad F, Ormezzano O, Vaisse B, Herpin D, Ribstein J, Bouhanick B, Mourad JJ, Ferrari E, Chatellier G, Sapoval M, Azarine A, Azizi M; DENERHTN Investigators. J Am Heart Assoc. 2017 Oct 10;6(10).
- 4. Twenty-Four-Hour Blood Pressure Monitoring to Predict and Assess Impact of Renal Denervation: The DENERHTN Study (Renal Denervation for Hypertension). Gosse P, Cremer A, Pereira H, Bobrie G, Chatellier G, Chamontin B, Courand PY, Delsart P, Denolle T, Dourmap C, Ferrari E, Girerd X, Michel Halimi J, Herpin D, Lantelme P, Monge M, Mounier-Vehier C, Mourad JJ, Ormezzano O, Ribstein J, Rossignol P, Sapoval M, Vaïsse B, Zannad F, Azizi M. Hypertension. 2017 Mar;69(3):494-500.
- Clinic Versus Ambulatory Blood Pressure in Resistant Hypertension: Impact of Antihypertensive Medication Nonadherence. A Post Hoc Analysis the DENERHTN Study. Hamdidouche I, Gosse P, Cremer A, Lorthioir A, Delsart P, Courand PY, Denolle T, Halimi JM, Girerd X, Ormezzano O, Rossignol P, Pereira P, Azizi M; DENERHTN Investigators. Hypertension. 2019 Nov;74(5):1096-1103.
- 6. Position Paper on the Role of Renal Denervation in the Management of the Difficult-to-Treat Hypertensive Patient. High Blood Press Cardiovasc Prev. Bruno RM, Taddei S, Borghi C, et al. Italian Society of Arterial Hypertension (SIIA) 2020;27(2):109-117.
- 7. Renal Denervation in Asia: Consensus Statement of the Asia Renal Denervation Consortium. Kario K, Kim BK, Aoki J, et al. Hypertension. 2020;75(3):590-602.
- 8. Device-based therapies for arterial hypertension. Lauder L, Azizi M, Kirtane AJ, Böhm M, Mahfoud F. Nat Rev Cardiol. 2020 Oct;17(10):614-628.
- 9. Rationale and design of two randomized sham-controlled trials of catheter-based renal denervation in subjects with uncontrolled hypertension in the absence (SPYRAL HTN-OFF MED Pivotal) and presence (SPYRAL HTN-ON MED Expansion) of antihypertensive medications: a novel approach using Bayesian design. Böhm M, Townsend RR, Kario K, et al. Clin Res Cardiol 2020; 109: 289–302.
- 10. Changes in 24-hour patterns of blood pressure in hypertension following renal denervation therapy. Kario K, Weber MA, Mahfoud F, et al. Hypertension 2019: 74: 244–49.
- 11. REDUCE HTN: REINFORCE. A randomized, sham-controlled trial of bipolar radiofrequency renal denervation for the treatment of hypertension. Weber MA, Kirtane AJ, Weir MR, et al. JACC CardiovascInterv 2020; 13: 461–70.
- 12. Renal denervation in patients with end-stage renal disease and resistant hypertension on long-term haemodialysis. Scalise F, Sole A, Singh G, Sorropago A et al. J Hypertens. 2020 May;38(5):936-942



13. Effect of renal denervation on blood pressure in the presence of antihypertensive drugs: 6-month efficacy and safety results from the SPYRAL HTN-ON MED proof-of-concept randomised trial. Kandzari DE, Böhm M, Mahfoud F, et al. Lancet 2018; 391: 2346–55.

14. Catheter-based renal denervation in patients with uncontrolled hypertension in the absence of antihypertensive medications (SPYRAL HTN-OFF MED): a randomised, sham-controlled, proof-of-concept trial. Townsend RR, Mahfoud F, Kandzari DE, et al. Lancet 2017; 390: 2160–70.